CLINICAL TRIAL: NCT05080777
Title: Pilot Pragmatic Clinical Trial to Embed Tele-Savvy Into Health Care Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Fortinsky, Richard, Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: U21-139-2
Record Dates: First submitted 2021-10-11; First posted 2021-10-18 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurocognitive Disorders; Neurodegenerative Diseases; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurocognitive Disorders; Neurodegenerative Diseases; Mental Disorders

STUDY DESIGN:
Intervention Model Description: Three Tele-Savvy programs, with 10 caregivers in each Tele-Savvy program cohort, will be held sequentially at each health care system site, for a total of 60 caregivers in 6 Tele-Savvy cohorts. Recruitment will occur in three waves, whereby caregivers will be randomly assigned at a 3:2 ratio to either Tele-Savvy or the attention control group until the first Tele-Savvy cohort is filled (first wave), followed by the same randomization procedure until the second and third Tele-Savvy cohorts are filled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-Savvy Group (Experimental): The participants will be enrolled into the Tele-Savvy group. Software analytics monitor caregivers' use of asynchronous material each week.
  Interventions: Behavioral: Tele-Savvy
- Attention Control Group (Active Comparator): The participants will be enrolled in the Caregiving During Crisis program. Software analytics monitor caregivers' use of asynchronous material each week.
  Interventions: Behavioral: Caregiving During Crisis (Educational Program)

INTERVENTIONS:
Behavioral: Tele-Savvy — A low-risk, psychoeducational, group-based intervention, is grounded in social learning and stress process theory and its main goal is to produce improved caregiver mastery over the symptom management skills commonly encountered when supervising and caring at home for an older adult living with ADRD. Over the 7-week program, there are synchronous and asynchronous activities each week. The synchronous portion includes weekly scheduled videoconferences (60-80 min) that serve as an online classroom in which facilitators lead lectures and discussions. Daily, caregivers access online 6- to 15-min prerecorded videos, each focused on one main learning objective. Caregivers can watch the lessons whenever and as often as they wish.
  Arms: Tele-Savvy Group
Behavioral: Caregiving During Crisis (Educational Program) — The attention control group will receive the self-guided Caregiving During Crisis program. Caregiving During Crisis is a fully online, asynchronous, professionally designed continuing education course aimed at developing the competency of informal caregivers of community-dwelling persons living with dementia to ensure the safety of that person and themselves during this time of the COVID-19 pandemic. The course, readily accessible by home computer or smartphone, describes methods of home infection control and prevention to create a Safe Home space, strategies for safely leaving and re-entering the home (e.g., to shop), additional strategies for safely allowing service personnel (e.g., home health aides or electricians) and select family members to enter the Safe Home space, and risk management strategies to frame decisions when/if COVID restrictions are relaxed or revoked.
  Arms: Attention Control Group

SUMMARY:
This cluster randomized pragmatic clinical trial will test the effectiveness and feasibility of embedding the Tele-Savvy intervention, a psychoeducational program for family and other informal caregivers of older adults living in the community with Alzheimer's disease and related dementia (ADRD), in two health care systems/clinical sites: UConn Health in Farmington, Connecticut, and Emory Healthcare in Atlanta, Georgia.

DETAILED DESCRIPTION:
This cluster randomized pragmatic clinical trial will test the effectiveness and feasibility of embedding the Tele-Savvy intervention, a psychoeducational program for family and other informal caregivers of older adults living in the community with Alzheimer's disease and related dementia (ADRD), in two health care systems/clinical sites: UConn Health in Farmington, Connecticut, and Emory Healthcare in Atlanta, Georgia. A total of 100 caregivers, 50 at each study site, will participate in this pilot study. At each site, 30 caregivers will be randomly assigned to receive the Tele-Savvy intervention, and 20 caregivers will be randomly assigned to receive the self-guided Caregiving During Crisis online program.

All 100 caregivers will complete identical self-administered questionnaires to measure the caregiver-specific outcome measures in this pilot study. Outcome measures will include caregiver mastery (primary outcome), caregiver response to specific memory and behavioral problems, and caregiver stress. Also, we will employ process measures of participation and engagement in the interventions for caregivers in both arms of the trial, as well as implementation outcomes via surveys with clinicians and Information Technology staff at each of the two clinical sites responsible for programming electronic medical records to enable capture and storage of caregiver outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Identified by EHR systems and confirmed by a health care provider as a family member or unpaid significant other who provides care at home for an older adult (age 65 or older) living with ADRD
* English speaking
* Able to understand study procedures and comply with them for the entire length of the study
* Access to appropriate video and audio technology to be able to participate in interventions

Exclusion Criteria:

* Unwilling to be randomized to receive either Tele-Savvy or Caregiving During Crisis
* Planning to admit the person living with ADRD to a nursing home on a long-term basis within 6 months of randomization.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard H. Fortinsky, PhD, Principal Investigator — UConn Health
Locations (2):
- United States (2):
  - UConn Health (Geriatrics Associates), Farmington, Connecticut
  - Emory HealthCare (IMCC), Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tele-Savvy Group | Attention Control Group
Started | 44 | 30
Completed | 26 (Based on number completed 3 month follow-up self-administered questionnaire.) | 10 (Based on number completed 3 month follow-up self-administered questionnaire.)
Not Completed | 18 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-Savvy Group | Attention Control Group | Total
Number analyzed (Participants) | 44 | 30 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (12.1) | 63.7 (11.2) | 65.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 22 | 54
  Male | 12 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 30 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 6 | 7 | 13
  White | 38 | 21 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 44 | 30 | 74
Marital Status [Count of Participants; unit: Participants]
  Married | 35 | 23 | 58
  Not Married | 9 | 7 | 16
Educational level [Count of Participants; unit: Participants]
  High school or some college | 7 | 6 | 13
  College degree | 15 | 11 | 26
  Graduate degree | 22 | 13 | 35
Relationship to person with dementia [Count of Participants; unit: Participants]
  Spouse/partner | 26 | 13 | 39
  Daughter | 13 | 11 | 24
  Son | 3 | 4 | 7
  Sibling | 1 | 1 | 2
  Other family member | 1 | 0 | 1
  Unknown | 0 | 1 | 1
Employed for pay outside the home [Count of Participants; unit: Participants]
  No | 30 | 22 | 52
  Yes | 14 | 8 | 22
Difficulty paying for basic needs [Count of Participants; unit: Participants]
  Not difficult at all | 32 | 17 | 49
  Not very difficult, somewhat or very difficult | 12 | 13 | 25
Primary caregiver [Count of Participants; unit: Participants]
  Yes | 36 | 27 | 63
  No | 8 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Caregiver Mastery
Description: Caregiving competence scale, minimum and maximum values 4-16, higher scores mean greater mastery.
Time Frame: pre-randomization; 3 months post-randomization; and 6 months post-randomization (6 months post-randomization for Emory site only)
Population: In the Tele-Savvy group, 40 participants had baseline data, 24 participants had 3-month follow-up data, and 16 participants had 6-month follow-up data. In the Attention Control group, 28 participants had baseline data, 10 participants had 3-month follow-up data, and 8 participants had 6-month follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group
Number analyzed (Participants) | 40 | 28
score on a scale
  Scores at baseline | 10.9 (2.1) | 11.5 (2.0)
  Scores at 3-month follow-up: number analyzed (Participants) | 24 | 10
  Scores at 3-month follow-up | 12.4 (2.0) | 12.0 (2.0)
  Scores at 6-month follow-up: number analyzed (Participants) | 16 | 8
  Scores at 6-month follow-up | 12.7 (1.3) | 12.8 (2.7)
Statistical Analysis 1: Comparison: Tele-Savvy Group vs Attention Control Group; Null hypothesis was that there would be no group differences, no time differences, and no group x time differences, in changes over time between the two treatment groups. Because this was a pilot and feasibility study, no power calculations were conducted; Test type: Equivalence — Group, Time, and Group x Time effect tests were performed using MLM; p = 0.295, Multilevel modeling (MLM) — .P-value shown is based on the Group x Time F statistic used in multilevel modeling (MLM)

2. Secondary Outcome: Change in Caregiver Reactions
Description: The reactions caregivers have to the behavioral and psychological symptoms expressed by persons living with dementia, were assessed using the Revised Memory and Behavior Problem Checklist (RMBPC). The RMBPC is a 24-item scale capturing caregiver reactions to 24 memory and behavior problems. Scores are computed based on the presence or absence of each problem first, and then for caregiver "reaction" or the extent to which caregivers were "bothered" or "upset" by each endorsed behavior. Reactions are assessed by asking how "upsetting" each behavior is to the caregiver on a Likert scale of 0 to 4 (0 = Not at all, 1= a little, 2 = moderately, 3 = very much, and 4 =extremely). Scores on the scale can range from 0-96, with higher scores meaning a worse outcome.
Time Frame: as for outcome 1
Population: In the Tele-Savvy group, 43 participants had baseline data, 26 participants had 3-month follow-up data, and 14 participants had 6-month follow-up data. In the Attention Control group, 29 participants had baseline data, 10 participants had 3-month follow-up data, and 8 participants had 6-month follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group
Number analyzed (Participants) | 43 | 29
score on a scale
  Scores at baseline | 22.4 (10.9) | 19.4 (12.3)
  Scores at 3-month follow-up: number analyzed (Participants) | 26 | 10
  Scores at 3-month follow-up | 17.6 (12.2) | 9.4 (13.0)
  Scores at 6-month follow-up: number analyzed (Participants) | 14 | 8
  Scores at 6-month follow-up | 17.2 (8.7) | 10.1 (7.3)
Statistical Analysis 1: Comparison: Tele-Savvy Group vs Attention Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Group, time, and group x time effect tests were performed using multilevel modeling (MLM); p = 0.570, MLM — P-value shown is based on the group x time F statistic used in MLM

3. Secondary Outcome: Change in Caregiver Stress
Description: The Perceived Stress Scale (PSS) is a 14-item instrument designed to measure the degree to which situations in one's life are appraised as stressful. Higher score reflects higher perceived stress. PSS items were designed to tap the degree to which respondents found their lives unpredictable, uncontrollable, and overloading. The scale also includes a number of direct queries about current levels of experienced stress. Each item is scored from 0 (never) to 4 (very often), for a possible score range of 0-56, with higher scores meaning worse outcomes.
Time Frame: pre-randomization; 3 months post-randomization; and 6 months post-randomization (6-month post randomization for Emory site only)
Population: In the Tele-Savvy group, 44 participants had baseline data, 26 participants had 3-month follow-up data, and 15 participants had 6-month follow-up data. In the Attention Control group, 30 participants had baseline data, 10 participants had 3-month follow-up data, and 8 participants had 6-month follow-up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tele-Savvy Group | Attention Control Group
Number analyzed (Participants) | 44 | 30
score on a scale
  Scores at baseline | 25.6 (6.6) | 24.5 (9.5)
  Scores at 3-month follow-up: number analyzed (Participants) | 26 | 10
  Scores at 3-month follow-up | 21.1 (5.5) | 15.2 (7.3)
  Scores at 6-month follow-up: number analyzed (Participants) | 15 | 8
  Scores at 6-month follow-up | 19.9 (5.7) | 16.8 (9.2)
Statistical Analysis 1: Comparison: Tele-Savvy Group vs Attention Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Group, time, and time x group effect tests were performed using multilevel modeling (MLM); p = 0.461, MLM — P-value shown is based on the group x time F statistic used in MLM

ADVERSE EVENTS:
Time Frame: In this pragmatic clinical trial testing an education and support intervention, adverse event occurrence was monitored during the 7-week duration of the intervention period for each caregiver.
Description: No differences in definitions between this study and the clinicaltrials.gov definitions.
Arm/Group | Tele-Savvy Group | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/30
Other Adverse Events (participants affected / at risk) | 0/44 | 0/30

LIMITATIONS AND CAVEATS:
Modest levels of outcome ascertainment at follow-up time points were due to the pragmatic nature of this pilot clinical trial, in which study participants (caregivers) received limited reminders from study personnel to submit follow-up self-administered questionnaires.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-12): https://cdn.clinicaltrials.gov/large-docs/77/NCT05080777/Prot_SAP_000.pdf